CLINICAL TRIAL: NCT00121264
Title: A Phase I Dose-Escalation Study of Intravenous 17-Allylaminogeldanamycin (17-AAG) [NSC 330507and Oral BAY 43-9006 [NSC 724772] Administered in Patients With Pretreated Advanced Solid Tumors
Brief Title: 17-AAG and Sorafenib in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03194; NCI-2012-03194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR434803; C-2890 (Other: Barbara Ann Karmanos Cancer Institute); 6972 (Other: CTEP); U01CA062487 (NIH); P30CA022453 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Sorafenib; tanespimycin; Magnetic Resonance Spectroscopy

ARMS (1):
- Treatment (sorafenib tosylate, tanespimycin) (Experimental): Patients receive oral sorafenib twice daily on days -14 to 28 in course 1 and on days 1-28 in all subsequent courses. Patients also receive 17-AAG IV over 3 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: tanespimycin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: magnetic resonance imaging

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: magnetic resonance imaging — Correlative studies
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-AAG when given together with sorafenib in treating patients with unresectable or metastatic solid tumors. Drugs used in chemotherapy, such as 17-AAG, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving 17-AAG together with sorafenib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To recommend a phase II dose for 17AAG (once weekly intravenously for 3 of 4 weeks), in combination with BAY 43-9006 (twice daily orally), by determining the feasibility, safety, dose limiting toxicities and the maximally tolerated dose.

SECONDARY OBJECTIVES:

I. To evaluate the modulation of pharmacodynamic effects and to investigate the interaction between the two mechanisms of action when used in combination by: Studying surrogate tissue and tumor cell signaling by Western blotting. Evaluating tumor blood flow utilizing dynamic contrast enhanced MRI.

II. To study any pharmacokinetic interactions between these two agents. III. To assess preliminary anti-tumor activity of this combination.

OUTLINE: This is an open-label, multicenter, dose-escalation study of 17-N-allylamino 17-demethoxygeldanamycin (17-AAG).

Patients receive oral sorafenib twice daily on days -14 to 28 in course 1 and on days 1-28 in all subsequent courses. Patients also receive 17-AAG IV over 3 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 5-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that which 2 of 6 patients experience dose-limiting toxicity.

After completion of study therapy, patients are followed for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Prior chemotherapy is allowed; patients may not have received chemotherapy for 4 weeks prior to the initiation of study treatment and must have full recovery from the acute effects of any prior chemotherapy; patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to initiation of study treatment
* Prior radiation therapy is allowed; patients must have completed radiation at least 4 weeks prior to initiation of study treatment; patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
* Prior treatment with biologic systemic therapies is permitted except for 17-AAG or Bay 43-9006 administration; prior experimental therapies (non FDA-approved agents) and immunotherapies are allowed; patients may not have received these therapies for 4 weeks prior to the initiation of study treatment and must have =< grade 2 residual toxicities from the effects of these therapies
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of > 12 weeks
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal; for patients with hepatic metastases, AST/ALT =< 5 x institutional upper limit of normal are permitted
* Creatinine =< 1.5 x institutional upper limit of normal OR
* Creatinine clearance >= 60 mL/min for patients with creatinine levels above 1.5 x institutional ULN
* Tumor evaluation studies such as CT scans/MRI/X-rays/PSA should be performed within 28 days of starting protocol therapy
* Patients are required to have DLCO of >= 60% on pretreatment pulmonary function tests with no symptomatic pulmonary disease
* Women of child-bearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy, biologic therapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from acute AEs due to agents administered more than 4 weeks earlier
* Patients who have received any other investigational agents within 28 days of study entry
* Patients may not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study except for medications that are prescribed for supportive care but potentially may have anticancer effect (i.e. megestrol acetate, dexamethasone, bisphosphonates); these medications must have been started at least 1 month prior to enrollment on study; in addition, men receiving treatment for prostate cancer will be maintained at castrate levels of testosterone by continuation of luteinizing- releasing hormone agonists
* Patients with egg allergy are excluded as 17-AAG is formulated in egg phospholipid
* Patients with known, symptomatic brain metastases should be excluded from this clinical trial; patients with stable or asymptomatic brain metastases are eligible but should not be taking enzyme-inducing anticonvulsants and should be maintained on stable steroid doses
* Patients with symptomatic pulmonary disease requiring medication including the following: dyspnea, dyspnea on exertion, paroxysmal nocturnal dyspnea, oxygen requirement and significant pulmonary disease, including chronic obstructive/restrictive pulmonary disease
* Patients that meet the Medicare criteria for home oxygen
* Patients with a prior history of chest radiation
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension (persistently elevated BP) or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and nursing women are excluded from this study
* HIV positive patients taking combination antiretroviral medications (HAART) would be excluded; HIV positive patients not being treated with anti-retroviral medications and otherwise meeting organ function criteria should be considered eligible
* Patients receiving CYP 3A4 inter active agent are eligible but should be studied carefully and where acceptable and appropriate substitutions of non-CYP interactive drugs should be undertaken; patients on therapeutic warfarin should be switched to LMW heparin; if appropriate a hematology consult should be obtained
* Patients with any impediment to swallowing tablets would be excluded
* Patients taking rifampin, St. John's wort and enzyme inducing anticonvulsant agents (e.g. phenytoin, phenobarbital) are excluded
* Patients with bleeding diathesis or patients taking oral anticoagulation with warfarin are excluded
* The use of concomitant medications that prolong or may prolong QTc are excluded
* Patients who have significant cardiac disease including heart failure that meet New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias, or poorly controlled angina are excluded
* Patients with a prior history of cardiac or pulmonary toxicity after receiving anthracyclines such as doxorubicin, daunorubicin, mitoxantrone, bleomycin or BCNU
* Patients with a greater or equal to grade 2 pulmonary or cardiac symptoms prior to study entry
* Patients who have a history of serious ventricular arrhythmia (VT or VF, >= 3 beats in a row), QTc> 450 msec for men and 470 msec for women, or LVEF =< 40% by MUGA are excluded
* Patients with a history of prior radiation that potentially included the heart in the field (e.g., mantle)
* Patients with active ischemic heart disease within 12 months
* Patients with a history of uncontrolled dysrhythmias or requiring antiarrythmic drugs; patients with congenital long QT syndrome
* Patients with left bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) based on the incidence of dose-limiting toxicity (DLT) as assessed by NCI CTCAE version 3.0 | 42 days
DLT as assessed by NCI CTCAE version 3.0 | 42 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters of sorafenib tosylate and tanespimycin | At baseline, at 0.5, 1, 2, 3, 4, 6, 9, and 12 hours of day 1, at 0.5, 1, and 2 hours on day 15, at 24 and 48 hours on days 16 and 17
  Descriptive PK studies will be performed for the combination to determine if there is any correlation with toxicity, efficacy or interaction. Plasma concentrations will be compared with in vitro and in vivo concentrations found to be effective in pre-clinical studies.
Pharmacodynamic effects of sorafenib tosylate and tanespimycin on surrogate markers and tumor tissue signaling by Western blotting | At baseline and at day -1, 14, and 18
Change in blood flow using dynamic contract enhanced MRI | At baseline, at days -3 to 1, and at days 15-22
Antitumor activity of this combination according to RECIST | Up to 60 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulka Vaishampayan, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States